CLINICAL TRIAL: NCT00275990
Title: AngioJET Rheolytic Thrombectomy Before Direct Infarct Artery STENTing in Patients Undergoing Primary PCI for Acute Myocardial Infarction: [JETSTENT] Study
Brief Title: AngioJET Thrombectomy and STENTing for Treatment of Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: JETSTENT
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Myocardial Infarction
Keywords: coronary thrombectomy; thrombectomy for acute myocardial infarction; C14.280.647.500; C14.907.553.355.500
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- thrombectomy before stenting (Experimental): thrombectomy before stenting
  Interventions: Device: rheolytic thrombectomy with direct stenting
- directing stenting alone (Active Comparator): directing stenting alone
  Interventions: Device: direct stenting

INTERVENTIONS:
Device: rheolytic thrombectomy with direct stenting
  Arms: thrombectomy before stenting
Device: direct stenting
  Arms: directing stenting alone

SUMMARY:
The purpose of this study is to determine whether prompt removal of thrombus (blood clot) from a blocked coronary artery using the AngioJet rheolytic thrombectomy device will result in improved blood flow within the heart and a smaller final infarct size (reduced injury to the heart muscle).

DETAILED DESCRIPTION:
Occlusive thrombosis triggered by a disrupted or eroded atherosclerotic plaque is the anatomic substrate of most acute myocardial infarctions (AMI). Macro- and microembolization of thrombus during percutaneous coronary intervention (PCI) in AMI is frequent and may result in obstruction of the microvessel network, and decreased efficacy of reperfusion and myocardial salvage. Direct stenting without predilation or postdilation is the most simplistic approach to the problem of embolization, and may decrease embolization and the incidence of the no-reflow phenomenon. Other approaches to the problem of microvessel embolization include percutaneous rheolytic thrombectomy (RT) with the AngioJet catheter before stent implantation. The objectives of the study are: to assess whether RT before direct infarct artery stenting results in improved reperfusion success in patients with acute ST-segment elevation myocardial infarction (STEMI) and angiographically evident thrombus; and to validate a technique for use of the AngioJet RT catheter in the treatment of STEMI.

Comparisons: Treatment with AngioJet RT immediately before direct infarct artery stenting versus direct stenting alone, in patients with STEMI and angiographically visible thrombus presenting within 6 hours of symptom onset for primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years
* ST-segment elevation myocardial infarction
* Angiographically visible thrombus
* Presentation within 6 hours of symptom onset for primary percutaneous coronary intervention
* Patient, or relative or legal guardian,provides written informed consent
* Patient has no childbearing potential or is not pregnant

Exclusion Criteria:

* Prior administration of thrombolysis for current MI
* Participation in another Study
* Major surgery within past 6 weeks
* History of stroke within 30 days, or any history of hemorrhagic stroke
* Severe hypertension (systolic BP > 200 mm Hg or diastolic BP > 110 mm Hg) not controlled on antihypertensive therapy
* Known neutropenia ( <1000 neutrophils per mm3) or known severe thrombocytopenia (< 50,000 platelets per mm3)
* Known prior history of renal insufficiency
* Co-morbidities with expected survival < 1 year
* Patient unwilling to receive blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
ST-segment resolution at 30 minutes post-PCI, assessed by 12-lead ECG | 30 minutes post procedure
Infarction size measured by technetium Tc 99m sestamibi imaging at 30 days | 30 days post-procedure

SECONDARY OUTCOMES:
Post-procedure- TIMI flow, TIMI myocardial blush, and corrected TIMI frame count | post-procedure
30 days- Technetium Tc 99m sestamibi infarct size, MACE | 30 days post-procedure
6 months- MACE | 6 months post-procedure
12 months- MACE | 12 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Antoniucci, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi, Florence, ITALY; Antonio Colombo, MD, Principal Investigator — San Raffaelle Hospital, Milan ITALY
Locations (1):
- Careggi Hospital, Division of Cardiology, Florence, Italy

REFERENCES:
- [Background] Antoniucci D, Valenti R, Migliorini A, Parodi G, Memisha G, Santoro GM, Sciagra R. Comparison of rheolytic thrombectomy before direct infarct artery stenting versus direct stenting alone in patients undergoing percutaneous coronary intervention for acute myocardial infarction. Am J Cardiol. 2004 Apr 15;93(8):1033-5. doi: 10.1016/j.amjcard.2004.01.011. PMID 15081450
- [Result] Migliorini A, Stabile A, Rodriguez AE, Gandolfo C, Rodriguez Granillo AM, Valenti R, Parodi G, Neumann FJ, Colombo A, Antoniucci D; JETSTENT Trial Investigators. Comparison of AngioJet rheolytic thrombectomy before direct infarct artery stenting with direct stenting alone in patients with acute myocardial infarction. The JETSTENT trial. J Am Coll Cardiol. 2010 Oct 12;56(16):1298-306. doi: 10.1016/j.jacc.2010.06.011. Epub 2010 Aug 5. PMID 20691553